CLINICAL TRIAL: NCT07235319
Title: A Multicenter, Open-Label, Randomized Phase III Non-Inferiority Trial of PD-1 Inhibitor Plus Chemotherapy Followed by Immediate Versus Salvage Locoregional Radiotherapy in De Novo Metastatic Nasopharyngeal Carcinoma
Brief Title: PD-1 Inhibitor Plus Chemotherapy Followed by Immediate Versus Salvage Locoregional Radiotherapy in De Novo Metastatic NPC
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Principal Investigator, Sun Yet-Sen University Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-FXY-252
Record Dates: First submitted 2025-11-13; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Nasopharangeal Cancer; Distant Metastasis
Keywords: Locoregional radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate locoregional radiotherapy group (Active Comparator): Immediate locoregional radiotherapy
  Interventions: Radiation: Immediate locoregional radiotherapy
- Salvage locoregional radiotherapy group (Experimental): Salvage locoregional radiotherapy
  Interventions: Radiation: Salvage locoregional radiotherapy

INTERVENTIONS:
Radiation: Immediate locoregional radiotherapy — Immediate locoregional radiotherapy (LRRT) with concurrent chemotherapy + PD-1 inhibitor Maintenance.
  Concurrent chemotherapy:
  Cisplatin (DDP) 80mg/m², starting on day 1 of radiotherapy, administered every 3 weeks during radiotherapy for a total of 3 cycles.
  PD-1 inhibitor maintenance therapy:
  Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  Arms: Immediate locoregional radiotherapy group
Radiation: Salvage locoregional radiotherapy — PD-1 inhibitor maintenance + Salvage locoregional radiotherapy
  PD-1 inhibitor maintenance therapy:Toripalimab 240 mg IV on day 1 every 3 weeks, or Tislelizumab 200 mg IV on day 1 every 3 weeks, or Camrelizumab 200 mg IV on day 1 every 3 weeks, continued until disease progression (per RECIST v1.1; if progression occurs in the nasopharynx or neck while metastatic lesions remain controlled, salvage locoregional radiotherapy* will be administered and PD-1 maintenance will continue until subsequent progression), unacceptable toxicity, patient withdrawal, or a maximum treatment duration of 2 years.
  *Concurrent chemotherapy: Cisplatin (DDP) 80 mg/m², starting on day 1 of radiotherapy, administered every 3 weeks during radiotherapy for a total of 3 cycles.
  Arms: Salvage locoregional radiotherapy group

SUMMARY:
This phase III randomized trial evaluates PD-1 inhibitor plus chemotherapy followed by immediate versus salvage locoregional radiotherapy in de novo metastatic nasopharyngeal carcinoma. The study aims to evaluate whether salvage locoregional radiotherapy is non-inferior to immediate radiotherapy following PD-1 inhibitor plus GP in de novo metastatic NPC, with potential for reduced toxicity.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is highly prevalent in Southern China, with approximately 15% of patients presenting with distant metastases at diagnosis. A PD-1 inhibitor combined with gemcitabine and cisplatin (GP) has become the standard first-line therapy for metastatic NPC. However, the survival benefit of adding immediate locoregional radiotherapy to PD-1 inhibitor plus GP in de novo metastatic NPC remains uncertain. This phase III randomized trial is designed to compare immediate versus salvage locoregional radiotherapy following PD-1 inhibitor plus GP in de novo metastatic NPC, with the objective of determining whether salvage radiotherapy is non-inferior to immediate radiotherapy while offering reduced toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 years, any gender.
2. Histologically confirmed differentiated non-keratinizing carcinoma or undifferentiated non-keratinizing carcinoma by tissue biopsy, with radiologically detectable metastatic lesions. Pathological confirmation of metastatic lesions is recommended but not mandatory.
3. ECOG performance status 0-1.
4. Stage IV NPC according to the 9th edition of the UICC/AJCC staging system.
5. No prior anti-tumor treatment for NPC (radiotherapy, chemotherapy, surgery, etc.).
6. Expected survival ≥ 3 months.
7. At least one measurable lesion per RECIST v1.1.
8. Achieved complete response (CR) or partial response (PR) after 4-6 cycles of chemotherapy plus PD-1 inhibitor therapy.
9. Adequate organ function within 14 days before first dose, defined as:

   Hematology：Hemoglobin ≥ 90 g/L，ANC ≥ 1.5 × 10⁹/L，Platelet count ≥ 100 × 10⁹/L Renal Function：Creatinine ≤ 1.5 × ULN, or creatinine clearance (CrCl) / eGFR ≥ 60 mL/min Liver Function：Total bilirubin ≤ 1.5 × ULN，AST and ALT ≤ 2.5 × ULN, or ≤ 5 × ULN in the presence of liver metastases
10. INR or PT ≤ 1.5 × ULN, unless on therapeutic anticoagulation and values within therapeutic range，aPTT ≤ 1.5 × ULN, unless on therapeutic anticoagulation and values within therapeutic range

Exclusion Criteria:

1. Prior anti-tumor therapy for nasopharyngeal carcinoma, including radiotherapy, chemotherapy, surgery, or immunotherapy.
2. Prior treatment with PD-1/PD-L1 or CTLA-4 inhibitors.
3. Presence of uncontrolled or symptomatic central nervous system (CNS) metastases.
4. History of other malignancies within the past 5 years, except adequately treated basal cell carcinoma, squamous cell skin cancer, or in-situ cervical cancer.
5. Active autoimmune disease or history of autoimmune disease requiring systemic treatment (e.g., corticosteroids, immunosuppressants) within the past 2 years, except for stable hypothyroidism, type 1 diabetes mellitus, or resolved childhood asthma/atopy.
6. Known history of active pulmonary tuberculosis (TB). Suspected active TB must be excluded by chest X-ray, sputum examination, and assessment of clinical signs and symptoms.
7. Hepatitis B: HBsAg positive with peripheral blood HBV DNA ≥ 1000 copies/mL
8. Hepatitis C: HCV antibody positive, eligible only if HCV RNA is negative
9. HIV infection
10. Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, unstable angina, myocardial infarction within 6 months, congestive heart failure ≥ NYHA class II, or serious arrhythmia).
11. Interstitial lung disease, non-infectious pneumonitis, or history of ≥ grade 2 pneumonitis.
12. Major surgery within 4 weeks before enrollment, or unhealed surgical wound.
13. Pregnant or breastfeeding women, or those planning pregnancy during the study period.
14. Known allergy or hypersensitivity to study drugs or their excipients.
15. Any condition that, in the investigator's judgment, would interfere with trial participation or interpretation of results.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2025-11-20 (Estimated); Primary Completion 2031-11-20 (Estimated); Study Completion 2034-11-20 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 year
  Defined as the time from random assignment to death from any cause.

SECONDARY OUTCOMES:
Locoregional progression-free survival | 2 year
  Defined as the time from random assignment to the occurrence of a locoregional progression.
Distant progression-free survival | 2 year
  Defined as the time from random assignment to the occurrence of a distant progression.
Progression free-survival | 2 year
  Defined as the time from random assignment to locoregional or distant progression, or death from any cause.
Incidence of Acute and Late Toxicity | 2 year
  Incidence of acute toxicity is calculated for each adverse event respectively and severity is evaluated on basis of Common Terminology Criteria for Adverse Events (CTCAE) 5.0 criteria. Late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
Quality of life (QoL) | 1 year
  The change of QoL from randomization to 1month, 3 months, 6 months and 1 year randomization. Assessed using the EORTC QoL questionnaire-C30 (EORTC QLQ-C30) version 3.0. This questionnaire comprises 30 questions, 24 aggregated into nine multi-question scales: five functioning scales (e.g., physical), three symptom scales (e.g., fatigue), and one global health status scale. The remaining six single-question (e.g., dyspnoea) scales assess symptoms. These 15 scales will be scored according to the official Scoring Manual of EORTC QLQ-C30.
Quality of life (QoL) | 1 year
  The change of QoL from randomization to 1month, 3 months, 6 months and 1 year randomization.QoL scores were assessed by using EORTC quality of life questionnaire(QLQ) Head and Neck. The QLQ-H&N35 is composed of seven multi-item symptom scales (pain, swallowing, sensation, speech, eating from a social,perspective, social interactions, and sexuality) and 11 single-item symptom scales (teeth, opening mouth,dry mouth, sticky saliva,coughing, felt ill, pain medication use, nutritional supplementation, feeding tube requirement, weight loss, and weight gain). All of the scales and items ranged in score from 0 to 100. A high score for a functional or global QoL scale represents a relatively high/healthy level of functional or global QoL, whereas a high score for a symptom scale or item represents a high number of symptoms or problems.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Hunan Cancer Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Guangxi Medical University Cancer Hospital, Nanning

IPD SHARING:
Plan to Share IPD: No